CLINICAL TRIAL: NCT00065065
Title: A Randomized, Placebo-controlled Trial of Rosiglitazone for Treatment of Ulcerative Colitis
Brief Title: A Trial of Rosiglitazone for Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Lewis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, James Lewis, Professor of Medicine and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROSIE; R01DK059961 (NIH)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Rosiglitazone; Ulcerative; Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Ulcer; Colitis | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosiglitazone (Experimental): 4 mg of rosiglitazone taken twice daily for 12 weeks.
  Interventions: Drug: Rosiglitazone
- placebo (Placebo Comparator): Identical in appearance to study drug taken twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — 4mg orally twice daily for 12 weeks
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Placebo — pill that looks identical to rosiglitazone
  Arms: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study evaluating rosiglitazone: 4 mg tablets or placebo tablets administered orally twice daily for 12 weeks. The purpose of the study is to evaluate the efficacy and safety of rosiglitazone in the treatment of mild to moderately active ulcerative colitis. Disease activity will be measured using a standard disease activity index. Calculation of the index requires patients to undergo flexible sigmoidoscopy at the start of the study and at week 12.

DETAILED DESCRIPTION:
Ulcerative colitis is a disease characterized by inflammation (the changes that happen when tissues in the body are injured) of all or a portion of the large intestine. There is presently no medical cure for ulcerative colitis, although surgical removal of the colon would cure the disease. Ulcerative colitis is generally treated with medications against diarrhea and infection, medications which suppress the immune system (the body system that protects a person against foreign substances) or with surgery.

It is thought that the chronic inflammation associated with ulcerative colitis may be related to the release of certain chemicals produced by the body. Rosiglitazone has been shown to inhibit the production of some of these chemicals. The active component of rosiglitazone has also been shown to improve colitis in animal models of colitis. The purpose of this study is to evaluate the benefit of the drug for ulcerative colitis by comparing it to placebo.

This is a randomized controlled trial of rosiglitazone versus placebo in patients who have failed to respond to 5-ASA therapy. Participants will be randomized to receive either rosiglitazone 4mg bid or placebo bid twice daily for a total of 12 weeks. Disease activity will be measured using the Disease Activity Index (DAI) at visits 3 through 8. Additional outcomes measured will include histological disease activity (visits 3 and 7) and quality of life using the IBDQ (visits 3 through 8). The principle analyses will be an intent-to-treat analysis to examine the efficacy of rosiglitazone at a dose of 4mg twice daily compared to placebo to achieve a partial or complete response. Additionally, the change in NF-κB activation prior to and following therapy with either placebo or rosiglitazone will be examined using immunohistochemistry techniques.

ELIGIBILITY:
INCLUSION CRITERIA: Participants must meet the following criteria for inclusion in the trial:

* Must sign and date the informed consent form
* At least 18 years of age
* Documented diagnosis (endoscopic, surgical or x-ray) of ulcerative colitis (UC)
* Mild to moderate ulcerative colitis indicated by Disease Activity Index score of greater than or equal to 4 and less than or equal to 10
* Unless the patient is intolerant of oral 5-ASA therapy, patient must be treated with a minimum of 2 gm daily of an oral 5-ASA agent for a minimum of 4 weeks during the current exacerbation of ulcerative colitis or immediately prior to study entry
* If treated with oral corticosteroids, dose must not exceed 20 mg per day of Prednisone or equivalent
* If treated with corticosteroids, dose must be stable for 4 weeks prior to study entry and remain on same dose throughout
* If treated with 6-mercaptopurine or azathioprine, must have been on medication for 4 months and a stable dose for 2 months prior to study entry
* If a female of childbearing age, the participant must have a negative serum pregnancy test and have been using a medically approved form of contraceptive birth control for 3 months prior to enrollment. Participants, both male and female, must also be willing to use medically approved contraceptive birth control (at least one barrier method) throughout the study
* If treated with rectal therapy, dose must be stable for 2 weeks prior to study entry and remain on same dose throughout

EXCLUSION CRITERIA: Participants will be ineligible for participation in the trial if they meet any of the following criteria:

* Severe ulcerative colitis indicated by Disease Activity Index score of greater than 10
* Class III or IV congestive heart failure by NYHA classification system
* Allergy to thiazolidinediones
* Presence of any medical condition with an expected survival of less than 1 year
* Participants receiving therapy with cyclosporin, anti-TNF therapy, or methotrexate within the last 2 months of screening
* Positive stool culture for enteric pathogens (salmonella, shigella, and campylobacter), positive C.difficile toxin, or positive stool ova and parasite exam
* Positive proteinuria by urine dipstick
* History of chronic liver disease or baseline liver chemistries greater than the upper limit of normal
* Diabetes mellitus requiring hypoglycemic agents
* Participation in study of experimental therapy within 2 months of first screening visit
* Has any of the following laboratory abnormalities: WBC < 3,000 per uL, Neutrophil < 1,000 cell/cu.mm, Platelets <75,000 per uL, INR > 1.2
* Participant is female and is pregnant or currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2002-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Study Director — University of Pennsylvania
Locations (13):
- United States (13):
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - Metropolitan Gastroenterology Group Practice/Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Maryland Digestive Diseases Research, Laurel, Maryland
  - Capitol Gastroenterology Consultants, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Atlantic Gastroenterology Associates, Egg Harbor, New Jersey
  - Wake Research Associates, Raleigh, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Avamar Center for Endoscopy, Warren, Ohio
  - University of Pennsylvania - Presbyterian Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Lewis JD, Lichtenstein GR, Deren JJ, Sands BE, Hanauer SB, Katz JA, Lashner B, Present DH, Chuai S, Ellenberg JH, Nessel L, Wu GD; Rosiglitazone for Ulcerative Colitis Study Group. Rosiglitazone for active ulcerative colitis: a randomized placebo-controlled trial. Gastroenterology. 2008 Mar;134(3):688-95. doi: 10.1053/j.gastro.2007.12.012. Epub 2007 Dec 7. PMID 18325386
- [Derived] Lewis JD, Chuai S, Nessel L, Lichtenstein GR, Aberra FN, Ellenberg JH. Use of the noninvasive components of the Mayo score to assess clinical response in ulcerative colitis. Inflamm Bowel Dis. 2008 Dec;14(12):1660-6. doi: 10.1002/ibd.20520. PMID 18623174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 15 clinical centers between September 6, 2002 and January 11, 2006.
Groups:
- Rosiglitazone: rosiglitazone (Avandia): 4mg orally twice daily for 12 weeks
- Placebo: Placebo identical to study drug twice daily for 12 weeks
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 52 | 53
Completed | 42 | 33
Not Completed | 10 | 20
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lack of Efficacy | 4 | 11
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rosiglitazone: rosiglitazone (Avandia): 4mg orally twice daily
- Placebo: Identical in appearance to study drug taken twice a day
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [31 to 49] | 46 [34 to 55] | 43 [31 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 30 | 34 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 48 | 50 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 53 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of Signs and Symptoms of UC at 12 Weeks
Description: Mayo score decrease >=2 points adjusted for age and smoking status.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 52 | 53
participants | 23 | 12
Statistical Analysis 1: Comparison: Rosiglitazone; Test type: Superiority or Other; p = .005, Regression, Logistic; Odds Ratio (OR) = 4.0, 95% CI [1.5 to 10.5]

2. Secondary Outcome: Number of Participants With Clinical Remission at 12 Weeks
Description: Mayo Score <=2 at 12 weeks post intervention
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 52 | 53
participants | 9 | 1

3. Secondary Outcome: Number of Participants With Endoscopic Remission at 12 Weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 52 | 53
Participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/52 | 5/53
Other Adverse Events (participants affected / at risk) | 36/52 | 30/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=52) | Placebo (N=53)
Worsening colitis requiring hospitalization and/or colectomy (Gastrointestinal disorders) | 1 (1) | 4 (4)
Bleeding after sigmoidoscopy biopsy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone (N=52) | Placebo (N=53)
Edema (General disorders) | 9 | 1
Fatigue (General disorders) | 4 | 3
Fever (General disorders) | 3 | 2
Constitutional symptoms-other (General disorders) | 5 | 3
Dermatologic skin - other (Skin and subcutaneous tissue disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 4 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 7
Vomiting (Gastrointestinal disorders) | 3 | 2
Gastrointestinal - other (Gastrointestinal disorders) | 6 | 8
Infection (Infections and infestations) | 5 | 3
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 5 | 1
Abdominal pain and cramping (Gastrointestinal disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Chest pain (General disorders) | 3 | 1
Headache (Nervous system disorders) | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain - other (General disorders) | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Proteinuria (Renal and urinary disorders) | 3 | 3
Decrease in hemoglobin concentration by 2 g/dL (Investigations) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No